CLINICAL TRIAL: NCT01845441
Title: A Randomized, Controlled Trial on Dexmedetomidine for Providing Adequate Sedation and Preserved Neurologic Examination for Endovascular Treatment of Acute Ischemic Stroke or Cerebral Vasospasm.
Brief Title: Use of Dexmedetomidine in Acute Stroke and Cerebral Vasospasm Interventions
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The principal investigator left employment at the sponsoring Institution
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 09-11-10; GIA#PRE-10-1003 (Other Grant/Funding Number: Hospira, Inc)
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Stroke; Brain Ischemia; Vasospasm, Intracranial; Hemorrhage, Intracranial
Keywords: Dexmedetomidine; Endovascular procedure; Stroke; Vasospasm, intracranial; Conscious sedation
MeSH Terms: conditions — Stroke; Brain Ischemia; Vasospasm, Intracranial; Intracranial Hemorrhages | interventions — Dexmedetomidine; Fentanyl; Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine arm (Experimental): Precedex will be started after randomization/prior to catheterization and will be stopped at the end of the procedure. It will be used for an average of 90 minutes and will be used as a continuous intravenous infusion started at 0.3 mcg/kg/hour. If HR > 80 and BP > 120/70, a full loading dose (1.0 mcg/kg/hour) will be administered over 10 minutes. If HR is 60 - 80 or systolic BP is 90 - 120, or age > 65 years, a reduced loading dose of 0.5 mcg/kg will be given over 10 minutes. If no volume overload history, 500mL of colloid (hespan or albumin) will be bolused with 0.2mg of glycopyrrolate. Every 10 minutes, Precedex will be titrated by 0.1 mcg/kg/hour to achieve and maintain RASS of 0 to -1.
  Interventions: Drug: Dexmedetomidine
- Control arm (Active Comparator): Our usual standard of care is to attempt the intervention without sedation. As per attending physician discretion, Fentanyl (50mcg) and/or Midazolam (0.5 mg) intravenous boluses will be used to control aggressive patient movement that adversely affects the technical capacity of the procedure. The boluses will be repeated at interval of 10 minutes, as necessary. Control arm patients will receive a normal saline placebo drip for the purposes of ensuring patient assessor blindness.
  Interventions: Drug: Fentanyl; Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Precedex will be given to randomized subjects in thi study to evaluate its efficacy in maintaining optimal sedation and preserving neurological exam.
  Other Names: Precedex
  Arms: Dexmedetomidine arm
Drug: Fentanyl — Patients in the control arm will receive no medication or standard sedative drug for the interventional procedure.
  Other Names: Sublimaze; Fentora; Instanyl
  Arms: Control arm
Drug: Midazolam — Patients in the control arm will receive no medication or standard sedative drug for the interventional procedure.
  Other Names: Dormicum; Hypnovel; Versed
  Arms: Control arm

SUMMARY:
Dexmedetomidine is a unique sedative medication able to provide sedation without causing respiratory depression and maintaining neurological functions. Patients having an acute ischemic stroke and need to undergo endovascular therapy require constant assessment of their neurological status prior, during and after the interventional procedure. In this study the investigators will compare the efficacy of Dexmedetomidine to other standard sedative medications in providing optimal sedative effect while maintaining neurological function.

DETAILED DESCRIPTION:
Precedex is a unique FDA-approved intravenous medication for conscious sedation in that it allows for "arousable" sedation, which is particularly appealing for use in patients with compromised neurologic function. While Precedex has been shown to be equivalent, if not superior to, conventional sedation in the procedural setting, it has not yet been evaluated in the setting of endovascular treatment of acute stroke. This setting is particularly ripe for evaluation, as there is currently controversy over the best method for management of patient sedation in light of the auxiliary need to preserve neurologic function. In order to evaluate the benefit of Precedex in this setting, it must be compared to the usual standard of care. Through the investigators double blinded randomized trial, the investigators will obtain information on the comparison between two arms, one receiving Precedex and the other the usual standard of care at the investigators institution, for achieving and maintaining a pre-defined level of conscious sedation, while preserving baseline neurologic status. This assessment will optimistically serve as the basis for future large-scale studies and ultimately to the establishment of Precedex as a first-line sedative in the management of acute stroke and cerebral vasospasm patients undergoing endovascular intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke who require endovascular intervention with whom mNIHSS score can be obtained
* Patients with cerebral vasospasm suspiciousness with or without subarachnoid hemorrhage with whom mNIHSS score can be obtained.

Exclusion Criteria:

* History of severe hepatic disease or severe renal disease (GFR<20).
* Hemodynamic instability.
* Pregnancy.
* Known allergy to study drug.
* Evidence or history of cardiac electrophysiology instability including uncontrolled hemodynamically unstable complex atrial/ventricular arrhythmia or conduction block at the time of evaluation with the exception of atrial fibrillation, and heart rate less than 60 or systolic blood pressure less than 90.
* Respiratory compromise requiring intubation.
* Any medical (including history of cardiac conduction block, major hepatic or renal disease) or laboratory abnormality that may increase the risk associated with the trial participation or drug administration or may interfere with interpretation of trial results.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-04; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine A Blackham, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

REFERENCES:
- [Background] Arepally A, Oechsle D, Kirkwood S, Savader SJ. Safety of conscious sedation in interventional radiology. Cardiovasc Intervent Radiol. 2001 May-Jun;24(3):185-90. doi: 10.1007/s002700002549. PMID 11443407
- [Background] Penumbra Pivotal Stroke Trial Investigators. The penumbra pivotal stroke trial: safety and effectiveness of a new generation of mechanical devices for clot removal in intracranial large vessel occlusive disease. Stroke. 2009 Aug;40(8):2761-8. doi: 10.1161/STROKEAHA.108.544957. Epub 2009 Jul 9. PMID 19590057
- [Background] Smith WS, Sung G, Saver J, Budzik R, Duckwiler G, Liebeskind DS, Lutsep HL, Rymer MM, Higashida RT, Starkman S, Gobin YP; Multi MERCI Investigators; Frei D, Grobelny T, Hellinger F, Huddle D, Kidwell C, Koroshetz W, Marks M, Nesbit G, Silverman IE. Mechanical thrombectomy for acute ischemic stroke: final results of the Multi MERCI trial. Stroke. 2008 Apr;39(4):1205-12. doi: 10.1161/STROKEAHA.107.497115. Epub 2008 Feb 28. PMID 18309168
- [Background] Gupta R, Vora NA, Horowitz MB, Tayal AH, Hammer MD, Uchino K, Levy EI, Wechsler LR, Jovin TG. Multimodal reperfusion therapy for acute ischemic stroke: factors predicting vessel recanalization. Stroke. 2006 Apr;37(4):986-90. doi: 10.1161/01.STR.0000209303.02474.27. Epub 2006 Mar 9. PMID 16527997
- [Background] Furlan A, Higashida R, Wechsler L, Gent M, Rowley H, Kase C, Pessin M, Ahuja A, Callahan F, Clark WM, Silver F, Rivera F. Intra-arterial prourokinase for acute ischemic stroke. The PROACT II study: a randomized controlled trial. Prolyse in Acute Cerebral Thromboembolism. JAMA. 1999 Dec 1;282(21):2003-11. doi: 10.1001/jama.282.21.2003. PMID 10591382
- [Background] Flaherty ML, Woo D, Kissela B, Jauch E, Pancioli A, Carrozzella J, Spilker J, Sekar P, Broderick J, Tomsick T. Combined IV and intra-arterial thrombolysis for acute ischemic stroke. Neurology. 2005 Jan 25;64(2):386-8. doi: 10.1212/01.WNL.0000149529.78396.B0. PMID 15668451
- [Background] Haslam PJ, Yap B, Mueller PR, Lee MJ. Anesthesia practice and clinical trends in interventional radiology: a European survey. Cardiovasc Intervent Radiol. 2000 Jul-Aug;23(4):256-61. doi: 10.1007/s002700010065. PMID 10960537
- [Background] Abou-Chebl A, Lin R, Hussain MS, Jovin TG, Levy EI, Liebeskind DS, Yoo AJ, Hsu DP, Rymer MM, Tayal AH, Zaidat OO, Natarajan SK, Nogueira RG, Nanda A, Tian M, Hao Q, Kalia JS, Nguyen TN, Chen M, Gupta R. Conscious sedation versus general anesthesia during endovascular therapy for acute anterior circulation stroke: preliminary results from a retrospective, multicenter study. Stroke. 2010 Jun;41(6):1175-9. doi: 10.1161/STROKEAHA.109.574129. Epub 2010 Apr 15. PMID 20395617
- [Background] Varma MK, Price K, Jayakrishnan V, Manickam B, Kessell G. Anaesthetic considerations for interventional neuroradiology. Br J Anaesth. 2007 Jul;99(1):75-85. doi: 10.1093/bja/aem122. Epub 2007 Jun 11. PMID 17562678
- [Background] Chamczuk AJ, Ogilvy CS, Snyder KV, Ohta H, Siddiqui AH, Hopkins LN, Levy EI. Elective stenting for intracranial stenosis under conscious sedation. Neurosurgery. 2010 Nov;67(5):1189-93; discussion 1194. doi: 10.1227/NEU.0b013e3181efbcac. PMID 20871450
- [Background] Stoneburner JM, Nishanian GP, Cukingnan RA, Carey JS. Carotid endarterectomy using regional anesthesia: a benchmark for stenting. Am Surg. 2002 Dec;68(12):1120-3. PMID 12516822
- [Background] Hoffman WE, Kochs E, Werner C, Thomas C, Albrecht RF. Dexmedetomidine improves neurologic outcome from incomplete ischemia in the rat. Reversal by the alpha 2-adrenergic antagonist atipamezole. Anesthesiology. 1991 Aug;75(2):328-32. doi: 10.1097/00000542-199108000-00022. PMID 1677549
- [Background] Taiji K. [Dexmedetomidine hydrochloride (Precedex), a new sedative in intensive care, its pharmacological characteristics and clinical study result]. Nihon Yakurigaku Zasshi. 2004 Sep;124(3):171-9. doi: 10.1254/fpj.124.171. Japanese. PMID 15333990

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexmedetomidine Arm | Control Arm
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine Arm | Control Arm | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Patient Movements (Events) That Delay or Adversely Affect the Procedure Performance and Safety.
Description: Patient will be continuously monitored for movements that delays or adversely affect the performance of the procedure by the patient assessor in a safe and timely manner (an event). One minute interval between patient event assessments will be given to prevent subjective bias. After every one minute, it will be determined if an event has occurred. Over the length of the procedure, the total number of one-minute intervals with an event occurrence will be summed and then divided by the total of minutes in the procedure to obtain a standardized value as the primary outcome. This will allow for direct comparison of values across the procedures of varying length. This approach will be more systematic and more easily replicable than counting events directly, which requires interpretation as to when a movement event begins and ends, which can be difficult and more subjective.
Time Frame: Primary outcome will be assessed during the procedure, up to 4 hours.
Population: Data was not collected for one patient in the Dexmedetomidine arm.
Measure: Median (Standard Deviation); unit: Events
Arm/Group | Dexmedetomidine Arm | Control Arm
Number analyzed (Participants) | 3 | 3
Events | 30 (27.07397) | 36 (25.86503)

2. Secondary Outcome: Preserved Neurological Examination.
Description: Neurological status using modified NIHSS (National Institutes of Health Stroke Scale) is a 15-item neurologic examination stroke scale, between 0 and 4, with 0 being normal functioning and 4 being completely impaired.
Time Frame: Up to 8 hours
Population: Data not collected for one patient in the dexmedetomidine arm
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Dexmedetomidine Arm | Control Arm
Number analyzed (Participants) | 3 | 3
score on a scale | 19 (5.75) | 18.5 (2.250926)

3. Secondary Outcome: Maintenance of Optimal Sedation Target in Both Groups.
Description: Both arms will be assessed by the patient assessor with RASS score measurement at baseline and every 20 minutes thereafter for the length of the procedure (up to 8 hours) and then averaged together to get one over all score . In the Dexmedetomidine arm the drug will be titrated by 0.1mcg/Kg/hour by the treating physician clinical judgment, in order to achieve and maintain RASS of 0 - 1. In the control arm the drug adjustment will not be based on the RASS score, but by physician discretion only. It is a 10-point scale to determine sedation, with a score from +4 (very combative, violent, dangerous to staff) to -5 (unarousable, no response to voice or physical stimulation).
Time Frame: Up to 8 hours
Population: Data not collected for one patient on Dexmedetomidine arm.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Dexmedetomidine Arm | Control Arm
Number analyzed (Participants) | 3 | 3
score on a scale | -1 (2.417882) | 0 (1.7754)

ADVERSE EVENTS:
Time Frame: Up to 8 hours
Arm/Group | Dexmedetomidine Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT01845441/Prot_SAP_000.pdf